CLINICAL TRIAL: NCT02022930
Title: A Multi-center, Randomized, Double-blind Study to Evaluate the Safety and Efficacy of Hydros and Hydros-TA Joint Therapies for Management of Pain Associated With Osteoarthritis in the Knee
Brief Title: Hydros and Hydros-TA Joint Therapy for Pain Associated With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carbylan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR1.1
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydros (Experimental): Hydros Joint Therapy
  Interventions: Device: Hydros
- Hydros-TA (Experimental): Hydros-TA Joint Therapy
  Interventions: Device: Hydros-TA
- Triamcinolone acetonide (Active Comparator): Triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Device: Hydros
  Arms: Hydros
Device: Hydros-TA
  Arms: Hydros-TA
Drug: Triamcinolone Acetonide
  Arms: Triamcinolone acetonide

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Hydros-TA Joint Therapy for relief of pain due to OA of the knee. Hydros-TA is designed to provide fast acting and long lasting pain relief for up to six months with a single IA injection.

ELIGIBILITY:
Inclusion Criteria:

* Have radiographic evidence within the prior 6 months, as shown in the radiology reports, of OA grade 2 or 3 using Kellgren-Lawrence Grading for OA.
* Symptoms in the index knee for at least 12 months.
* Fully ambulatory Subject (ability to perform a 15 meters walk test).
* Male and female Subjects 40 through 85 years of age.

Exclusion Criteria:

* BMI >40 kg
* Secondary OA (acute knee injury, rheumatoid arthritis, gout, history of joint infection, osteonecrosis, chronic fibromyalgia) or other chronic autoimmune disease.
* Intra articular steroid therapy in last 3 months
* Intra articular viscosupplementation in last 6 months

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the WOMAC A subscale score for the treatment knee. | 2 weeks and 26 weeks

SECONDARY OUTCOMES:
Strict positive responders to treatment for symptomatic primary osteoarthritis of the knee | 26 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- St Leonards, New South Wales, Australia
- Canada (3):
  - London, Ontario
  - Oshawa
  - Québec
- Willemstad, Curacao, Netherlands Antilles